CLINICAL TRIAL: NCT05937373
Title: A Pilot Trial of Continuous Glucose Monitoring (CGM) Technology in Preoperative Assessment Clinic
Brief Title: Perioperative Continuous Glucose Monitoring
Acronym: CGM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of research funding support
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00097714
Record Dates: First submitted 2023-06-21; First posted 2023-07-10 (Actual); Results first posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2024-11

CONDITIONS: Diabetes Mellitus
Keywords: A1c; blood glucose changes; hyperglycemic and hypoglycemic events
MeSH Terms: conditions — Diabetes Mellitus | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Continuous Glucose Monitor (Experimental): CGM placed preoperative to monitor blood glucose and insulin correction to achieve perioperative glucose management
  Interventions: Device: Continuous Glucose monitor
- Standard of Care (Active Comparator): no study intervention-conventional glucose management per subjects medical providers as standard of care
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: Continuous Glucose monitor — Perioperative glucose management beginning preoperative through postoperative monitoring
  Arms: Continuous Glucose Monitor
Other: Standard of Care — no study intervention. participant follows current medical providers recommendations for glucose management
  Arms: Standard of Care

SUMMARY:
To evaluate use of continuous glucose monitoring (CGM) technology in the preoperative setting: evaluate feasibility of placement of CGM during preoperative clinic visit with intent to utilize CGM throughout perioperative period.

DETAILED DESCRIPTION:
To further study potential barriers related to loss of continuous glucose monitoring (CGM) data as it relates to use of electrocautery and grounding devices utilized in the perioperative setting. To assess how CGM technology could improve glycemic management in the perioperative setting, specifically in predicting and preventing hypoglycemic episodes as well as utilization for treating hyperglycemia with resultant improvement in patient morbidity, mortality, length of stay, and overall quality of life. CGM technology aids tremendously in data collection with recognition of glycemic patterns, as well as evaluating prediction of blood glucose changes including both hyperglycemic and hypoglycemic events. The availability of such a large volume of glycemic data has been shown to make a tremendous impact in patient care, resulting in statistically significant reductions in hemoglobin A1c, a decrease in hypoglycemia, a decrease in hospital admissions for diabetes complications, and improved overall quality of life and fear of hypoglycemia in patients using CGM technology.

ELIGIBILITY:
Inclusion Criteria:

* Participants that are 18 years of age or older with hyperglycemia and/or diabetes mellitus who will be undergoing surgery at Atrium Health Wake Forest Baptist
* smartphone compatible with Libre 2 phone application

Exclusion Criteria:

* Pregnant women will not be excluded from this study
* Participants undergoing surgery that would limit the placement of Continuous Glucose Monitoring (CGM) to the posterior aspect of the upper extremity will be excluded from this study
* neurosurgical type of surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-08-04 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Vishneski, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Continuous Glucose Monitor: Freestyle Libre 2 CGM placed preoperative to monitor blood glucose and insulin correction to achieve perioperative glucose management
- Standard of Care: No study intervention-conventional glucose management with Freestyle Libre Pro CGM per subjects medical providers as standard of care
Period: Overall Study
Arm/Group | Continuous Glucose Monitor | Standard of Care
Started | 11 | 11
Completed | 9 | 9
Not Completed | 2 | 2
Not completed — Out of Window | 2 | 0
Not completed — Device fell off prior to date of surgery | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuous Glucose Monitor | Standard of Care | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (5.67) | 62 (10.17) | 67 (9.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 6 | 9 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 11 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Disparities in Continuous Glucose Monitoring (CGM) Accuracy - Fingerstick Values
Description: Accuracy of CGM technology utilizing Dexcom G6 CGM and Freestyle Libre 2.0 CGM in the perioperative setting for glycemic management of patients with hyperglycemia and/or diabetes mellitus compared with current standard of care utilizing point of care blood glucose fingerstick Glucose values - Only Glucometers
Time Frame: Day 7
Measure: Mean (Standard Deviation); unit: Percentage of mmol/L
Units Other Than Participants: glucose values each group
Arm/Group | Continuous Glucose Monitor | Standard of Care
Number analyzed (Participants) | 9 | 9
Number analyzed (glucose values each group) | 67 | 99
Percentage of mmol/L | 4.32 (18.41) | 8.08 (37.73)

2. Primary Outcome: Disparities (Percentage Difference) in Continuous Glucose Monitoring (CGM) Accuracy - Comprehensive Metabolic Panel (CMP) / Basic Metabolic Panel (BMP)/ Blood Gas Values - Overall Number of Unit Analyzed (Glucose Values Each Group)
Description: Accuracy of CGM technology utilizing Dexcom G6 CGM and Freestyle Libre 2.0 CGM in the perioperative setting for glycemic management of patients with hyperglycemia and/or diabetes mellitus compared with current standard of care utilizing serum and arterial glucose values - Comprehensive Metabolic Panel (CMP) / Basic Metabolic Panel (BMP)/ blood gas values For each CMP/BMP/Blood Gas Value recorded in the Electronic Medical Record during the period of CGM wear, a percentage difference was calculated between the measured glucose value and the corresponding CGM value.
Time Frame: Day 7
Population: overall number of unit analyzed (glucose values each group)
Measure: Mean (Standard Deviation); unit: percent difference in blood glucose valu
Units Other Than Participants: unit analyzed - measured glucose value a
Arm/Group | Continuous Glucose Monitor | Standard of Care
Number analyzed (Participants) | 9 | 9
Number analyzed (unit analyzed - measured glucose value a) | 67 | 99
percent difference in blood glucose valu | 4.18 (15.86) | 1.20 (16.41)

3. Other Pre Specified Outcome: Patient Satisfaction Scores
Description: A patient satisfaction survey will be collected to further evaluate the patient's perspective of wearing a CGM in the perioperative period
Time Frame: Day 7
Population: VALUE NOT EVALUATED - Data not collected - patient satisfaction scores were not collected as a part of the data collection process
Arm/Group | Continuous Glucose Monitor | Standard of Care
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Percentage of Patients With Functioning Continuous Glucose Monitoring (CGM) - Arrived on Their Date of Surgery (DOS) With Working CGM
Description: Proportion of patients who present on day of surgery with CGM still in place and functioning
Time Frame: Day 7
Population: no study intervention-conventional glucose management per subjects medical providers as standard of care
  Standard of Care: no study intervention. participant follows current medical providers recommendations for glucose management
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Glucose Monitor | Standard of Care
Number analyzed (Participants) | 11 | 0
Participants | 9 | 0

5. Secondary Outcome: Disparities in Continuous Glucose Monitoring (CGM) Accuracy - Interference Amount
Description: Analysis of potential electrocautery interference in CGM data collection was performed through visual review of the CGM glucose data graphs for unexpected gaps or spikes during surgery. No such events were observed in the CGM outputs during the review. Disparities in CGM accuracy due to interference were reported as 0%.
Time Frame: Hour 24
Measure: Number; unit: Number of Discrepencies
Arm/Group | Continuous Glucose Monitor | Standard of Care
Number analyzed (Participants) | 9 | 9
Number of Discrepencies | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 7
Arm/Group | Continuous Glucose Monitor | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-07): https://cdn.clinicaltrials.gov/large-docs/73/NCT05937373/Prot_SAP_001.pdf
  • Informed Consent Form (2024-07-03): https://cdn.clinicaltrials.gov/large-docs/73/NCT05937373/ICF_000.pdf